CLINICAL TRIAL: NCT04308993
Title: Percutaneous Endoscopic Biliary Exploration in Complex Biliary Stone Disease: Cohort Study
Brief Title: Percutaneous Endoscopic Biliary Exploration in Complex Biliary Stone Disease
Status: Completed | Type: Observational
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Hanan Mesfer Alghamdi, Assistant professor of Surgery, Imam Abdulrahman Bin Faisal University
Other Study IDs: IAU-PEBE
Record Dates: First submitted 2020-03-06; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Biliary Stones
MeSH Terms: conditions — Cholecystolithiasis | interventions — Lithotripsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: percutaneous transhepatic choledochoscopy — percutaneous transhepatic choledochoscopy
  Other Names: extracorporeal shock wave lithotripsy (ESWL)

SUMMARY:
Patients with complex biliary stone disease are challenging to treat. The investigator present their experience in using urological interventions to treat challenging biliary stones.

Methods:

Fifteen patients with biliary calculi underwent 21 interventions using either extracorporeal shock wave lithotripsy (ESWL), percutaneous transhepatic choledochoscopy, percutaneous transcystic choledochoscopy, or a combination of these.

DETAILED DESCRIPTION:
The investigator conducted a retrospective review to investigate the outcomes of urological treatments for biliary calculi from January 1, 1999, to August 31, 2016, focusing on percutaneous endoscopic methods and/or ESWL. The primary outcomes of interest were symptom- and stone-free rates, length of hospital stay, and complications. Our institutional ethics review board approved the study (IRB-2018-01-119). Due to the retrospective nature of the study, the need for informed consent was waived. One endourologist evaluated all patients preoperatively.

Urological intervention techniques The three different approaches used (ESWL, PTHC, and PTCC) are described below.

ELIGIBILITY:
Inclusion Criteria:

* complete records

Exclusion Criteria:

* lost follow up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Most patients were elderly (median age, 60 years). The male-to-female ratio was higher than the norm for biliary stones (1:1.4). The most common reasons for failure of conventional endoscopic retrograde cholangiopancreatography (ERCP) were high American Society of Anesthesia (ASA) score (8 patients 53%), technical failure of ERCP (4 patients, 27%), previous Roux-en-Y gastric bypass (two patients, 13%), and post-common bile duct (CBD) injury with T-tube insertion (one patient, 7%). The stone sites were the CBD, gallbladder, and intrahepatic bile duct in nine (60%), three (20%), and three (20%) patients, respectively
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
symptoms | at least one year follow up
  success rate of biliary stone clearance or asymptomatic derbies

SECONDARY OUTCOMES:
ultrasound | one month
  evidence of stone clearance

OTHER OUTCOMES:
obstructive jaundice | one day
  biochemical evidence (Liver function test) of improvement

IPD SHARING:
Plan to Share IPD: Undecided